CLINICAL TRIAL: NCT02590068
Title: Effects of Chronic Viral Infection on Immune Response to Zoster Vaccination
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI at new institution and no further enrollment to take place.
Sponsor: Rockefeller University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OJE-0890; 5U19AI111825-02 (NIH)
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hepatitis C infected volunteers (Experimental): Zoster vaccine live (Zostavax), 0.65 ml dose, administered subcutaneously to Hepatitis C infected volunteers
  Interventions: Drug: Zoster vaccine live
- Healthy volunteers (Active Comparator): Zoster vaccine live (Zostavax), 0.65 ml dose, administered subcutaneously to healthy volunteers
  Interventions: Drug: Zoster vaccine live

INTERVENTIONS:
Drug: Zoster vaccine live — Single Zostavax vaccine, 0.65 ml dose, administered subcutaneously
  Other Names: Zostavax

SUMMARY:
This study aims to identify the innate and adaptive immune response to zoster vaccination. Half of the participants will be individuals with chronic hepatitis C, while the other half with healthy volunteers.The innate immune signature elicited by Zoster vaccination will be characterized by RNA-seq analysis of pre- and post-vaccination RNA from whole blood. We will compare fold changes in gene expression profiles pre- versus post-vaccination in each individual, as well as between the two arms of the study. RNA-seq will be used to assess innate immune activation by evaluating the changes to the expression levels of interferon-stimulated genes pre- and post-vaccination. Adaptive immune response will be determined by the traditional correlates of protection used in previous Zoster clinical studies in addition to flow cytometry24. Correlates of protection include antibody response, interferon gamma production and the frequency of responder cells post- vaccination24. For antibody production, we will perform Zoster glycoprotein ELISA (gpELISA) targeting IgG/IgM. The number and frequency of responder cells will be characterized by flow cytometry.

DETAILED DESCRIPTION:
Chronic HCV infection is associated with persistent innate immune activation and dampened cellular immune responses. Interferons (IFNs) are key mediators of the antiviral innate immune response, initiating the expression of interferon-stimulated genes (ISG) with numerous host protective effector functions. However, in chronic HCV, high pre-therapy expression of ISG and persistent activation of the innate immune system negatively predicts the response to IFN-based therapies and failure of viral clearance8. In addition, HCV persistence is also associated with HCV-specific-CD8+ T cell exhaustion. HCV-specific CD8+ T cell exhaustion is characterized by diminished ex vivo polyfunctionality, upregulation of negative costimulatory cell modulators and, decreased cellular proliferation and IFN production10,12. This phenotype is associated with the development of short-term effector CD8+ T cells rather than durable, long-term memory CD8+ T cells. Chronic bystander infections (e.g. chronic HCV), characterized by persistent inflammation have been linked to bystander (non-HCV specific) CD8+ T cell dysfunction. Bystander CD8+ T cell dysfunction significantly impairs the expansion of memory CD8+ T cells and could prevent the development of secondary immunological memory to new antigens and/or vaccines11,13. Clinically, chronic HCV has been associated with impaired immune response to Hepatitis B vaccination13,14,15. Only 40% to 60% of individuals with chronic HCV achieve seroprotective titers following HBV vaccination versus 90% to 95% in healthy subjects13,14. Specific immune defects responsible for HBV vaccine failure in HCV-infected patients are unknown at present. However, some studies have suggested that the blunting of the immune response to HBV vaccination is associated with lymphocyte dysfunction and upregulation of PD-1 expression on CD4+ T cells in HBV vaccine non-responders13,15.

In the United States, 99.5% of adults over 40 years have been infected with the Varicella zoster virus (VZV) and are at risk of Zoster virus reactivation (shingles) and its complications. Unilateral, painful, blistering rashes along dermatomes characterize shingles. Complications associated with shingles include acute or chronic pain, osteonecrosis, zoster ophthalmicus with visual impairment, increased risk of blindness and a 4-fold risk of cerebral vasculitis-associated stroke)1,2. Overall, complications of shingles have a negative impact on the quality of life and activities of daily living21,22. Zoster vaccine live (Zostavax®, Merck) is recommended for the prevention of shingles. Zoster vaccine is a live, attenuated vaccine that is licensed by the FDA for individuals older than 50 years without an underlying immune deficiency (HIV, malignancies, immunosuppression and transplantation). In non-immunocompromised individuals, Zoster vaccine decreases shingles by 51% in individuals between ages 60 - 89 years and 70% in individuals between 50 - 59 years of age. Chronic infections such as TB, malaria and chronic Hepatitis C virus (HCV) have been associated with increased susceptibility to other pathogens and decreased vaccination efficacy3-6. Although chronic HCV infection is not considered a clinically immunocompromised state, it is associated with persistent immune activation and decreased vaccination response7. Zostavax is routinely administered to chronic HCV patients. However, at present, no other study has documented the immune responses elicited by Zoster vaccination in this population. This study aims to identify the innate and adaptive immune signatures elicited by zoster vaccination in chronic HCV and healthy volunteers. Unrecognized suboptimal vaccine response in individuals with chronic immune dysregulated states (chronic bystander viral infections (HBV, HCV and HIV with CD4 >200), diabetes, advancing age, cancers and transplantation) could be potentially devastating and costly.

ELIGIBILITY:
Inclusion Criteria:

* Willing to receive the herpes zoster vaccine
* Volunteer chronically infected with HCV (as demonstrated by serology testing and have a viral load >1000 copies) without treatment
* Healthy volunteer without significant medical problems

Exclusion Criteria:

* Received any vaccine within a month prior to study vaccine
* Previous Zoster infection as an adult, >18 years
* HIV or Hepatitis B virus infection in the HCV and healthy arms
* For HCV-negative, healthy volunteers: History of HCV infection or positive HCV antibody test
* Participation in another clinical study of an investigational product currently or within the past 90 days, or expected particpation during this study
* In the opinion of the investigator, the volunteer is unlikely to comply with the study protocol
* Any clinically significant abnormality or medical history or physical examination including history of immunodeficiency or autoimmune disease (in addition to HCV infection, for HCV group)
* Currently taking systemic steroids or other immunomodulatory medications including anticancer medications and antiviral medications
* Any clinically significant acute or chronic medical condition requiring care by a primary care provider (e.g., diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that, in the opinion of the investigator, would preclude participation
* Male or female < 50 and > 70 years of age
* Is pregnant or lactating
* Clinical, laboratory, or biopsy evidence of cirrhosis
* Allergy to gelatin and/or neomycin
* ALT and/or AST > 3.5 times the ULN
* Immunosuppressed or immunodeficient individuals including those with a history of primary or acquired immunodeficiency states, leukemia, lymphoma or other malignant neoplasms affecting the bone marrow or lymphatic system and those on immunosuppressive therapy
* Individuals with active untreated tuberculosis
* Prior Varicella vaccination
* HCV volunteers who have a viral load of <1000 copies

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oyebisi Jegede, MBBS, PhD, Principal Investigator — The Rockefeller University Center for Clinical and Translational Studies
Locations (1):
- Rockefeller University Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oxman MN, Levin MJ, Johnson GR, Schmader KE, Straus SE, Gelb LD, Arbeit RD, Simberkoff MS, Gershon AA, Davis LE, Weinberg A, Boardman KD, Williams HM, Zhang JH, Peduzzi PN, Beisel CE, Morrison VA, Guatelli JC, Brooks PA, Kauffman CA, Pachucki CT, Neuzil KM, Betts RF, Wright PF, Griffin MR, Brunell P, Soto NE, Marques AR, Keay SK, Goodman RP, Cotton DJ, Gnann JW Jr, Loutit J, Holodniy M, Keitel WA, Crawford GE, Yeh SS, Lobo Z, Toney JF, Greenberg RN, Keller PM, Harbecke R, Hayward AR, Irwin MR, Kyriakides TC, Chan CY, Chan IS, Wang WW, Annunziato PW, Silber JL; Shingles Prevention Study Group. A vaccine to prevent herpes zoster and postherpetic neuralgia in older adults. N Engl J Med. 2005 Jun 2;352(22):2271-84. doi: 10.1056/NEJMoa051016. PMID 15930418
- [Background] Lin F, Hadler JL. Epidemiology of primary varicella and herpes zoster hospitalizations: the pre-varicella vaccine era. J Infect Dis. 2000 Jun;181(6):1897-905. doi: 10.1086/315492. Epub 2000 Jun 5. PMID 10837168
- [Background] Abu-Raddad LJ, Patnaik P, Kublin JG. Dual infection with HIV and malaria fuels the spread of both diseases in sub-Saharan Africa. Science. 2006 Dec 8;314(5805):1603-6. doi: 10.1126/science.1132338. PMID 17158329
- [Background] Zhu J, Hladik F, Woodward A, Klock A, Peng T, Johnston C, Remington M, Magaret A, Koelle DM, Wald A, Corey L. Persistence of HIV-1 receptor-positive cells after HSV-2 reactivation is a potential mechanism for increased HIV-1 acquisition. Nat Med. 2009 Aug;15(8):886-92. doi: 10.1038/nm.2006. Epub 2009 Aug 2. PMID 19648930
- [Background] Pisell TL, Hoffman IF, Jere CS, Ballard SB, Molyneux ME, Butera ST, Lawn SD. Immune activation and induction of HIV-1 replication within CD14 macrophages during acute Plasmodium falciparum malaria coinfection. AIDS. 2002 Jul 26;16(11):1503-9. doi: 10.1097/00002030-200207260-00007. PMID 12131188
- [Background] Bahgat MM, El-Far MA, Mesalam AA, Ismaeil AA, Ibrahim AA, Gewaid HE, Maghraby AS, Ali MA, Abd-Elshafy DN. Schistosoma mansoni soluble egg antigens enhance HCV replication in mammalian cells. J Infect Dev Ctries. 2010 May 1;4(4):226-34. doi: 10.3855/jidc.522. PMID 20440060
- [Background] Stelekati E, Wherry EJ. Chronic bystander infections and immunity to unrelated antigens. Cell Host Microbe. 2012 Oct 18;12(4):458-69. doi: 10.1016/j.chom.2012.10.001. PMID 23084915
- [Background] Schoggins JW, Wilson SJ, Panis M, Murphy MY, Jones CT, Bieniasz P, Rice CM. A diverse range of gene products are effectors of the type I interferon antiviral response. Nature. 2011 Apr 28;472(7344):481-5. doi: 10.1038/nature09907. Epub 2011 Apr 10. PMID 21478870
- [Background] Metz P, Dazert E, Ruggieri A, Mazur J, Kaderali L, Kaul A, Zeuge U, Windisch MP, Trippler M, Lohmann V, Binder M, Frese M, Bartenschlager R. Identification of type I and type II interferon-induced effectors controlling hepatitis C virus replication. Hepatology. 2012 Dec;56(6):2082-93. doi: 10.1002/hep.25908. Epub 2012 Oct 14. PMID 22711689
- [Background] Wherry EJ, Ha SJ, Kaech SM, Haining WN, Sarkar S, Kalia V, Subramaniam S, Blattman JN, Barber DL, Ahmed R. Molecular signature of CD8+ T cell exhaustion during chronic viral infection. Immunity. 2007 Oct;27(4):670-84. doi: 10.1016/j.immuni.2007.09.006. Epub 2007 Oct 18. PMID 17950003
- [Background] Stelekati E, Shin H, Doering TA, Dolfi DV, Ziegler CG, Beiting DP, Dawson L, Liboon J, Wolski D, Ali MA, Katsikis PD, Shen H, Roos DS, Haining WN, Lauer GM, Wherry EJ. Bystander chronic infection negatively impacts development of CD8(+) T cell memory. Immunity. 2014 May 15;40(5):801-13. doi: 10.1016/j.immuni.2014.04.010. PMID 24837104
- [Background] Urbani S, Amadei B, Tola D, Massari M, Schivazappa S, Missale G, Ferrari C. PD-1 expression in acute hepatitis C virus (HCV) infection is associated with HCV-specific CD8 exhaustion. J Virol. 2006 Nov;80(22):11398-403. doi: 10.1128/JVI.01177-06. Epub 2006 Sep 6. PMID 16956940
- [Background] Moorman JP, Zhang CL, Ni L, Ma CJ, Zhang Y, Wu XY, Thayer P, Islam TM, Borthwick T, Yao ZQ. Impaired hepatitis B vaccine responses during chronic hepatitis C infection: involvement of the PD-1 pathway in regulating CD4(+) T cell responses. Vaccine. 2011 Apr 12;29(17):3169-76. doi: 10.1016/j.vaccine.2011.02.052. Epub 2011 Mar 3. PMID 21376795
- [Background] Wiedmann M, Liebert UG, Oesen U, Porst H, Wiese M, Schroeder S, Halm U, Mossner J, Berr F. Decreased immunogenicity of recombinant hepatitis B vaccine in chronic hepatitis C. Hepatology. 2000 Jan;31(1):230-4. doi: 10.1002/hep.510310134. PMID 10613751
- [Background] Crawford A, Angelosanto JM, Kao C, Doering TA, Odorizzi PM, Barnett BE, Wherry EJ. Molecular and transcriptional basis of CD4(+) T cell dysfunction during chronic infection. Immunity. 2014 Feb 20;40(2):289-302. doi: 10.1016/j.immuni.2014.01.005. Epub 2014 Feb 13. PMID 24530057
- [Background] Maecker HT, McCoy JP, Nussenblatt R. Standardizing immunophenotyping for the Human Immunology Project. Nat Rev Immunol. 2012 Feb 17;12(3):191-200. doi: 10.1038/nri3158. PMID 22343568
- [Background] Levin MJ, Smith JG, Kaufhold RM, Barber D, Hayward AR, Chan CY, Chan IS, Li DJ, Wang W, Keller PM, Shaw A, Silber JL, Schlienger K, Chalikonda I, Vessey SJ, Caulfield MJ. Decline in varicella-zoster virus (VZV)-specific cell-mediated immunity with increasing age and boosting with a high-dose VZV vaccine. J Infect Dis. 2003 Nov 1;188(9):1336-44. doi: 10.1086/379048. Epub 2003 Oct 17. PMID 14593591
- [Background] Sauerbrei A, Wutzler P. Serological detection of varicella-zoster virus-specific immunoglobulin G by an enzyme-linked immunosorbent assay using glycoprotein antigen. J Clin Microbiol. 2006 Sep;44(9):3094-7. doi: 10.1128/JCM.00719-06. PMID 16954232
- [Background] Soneson C, Delorenzi M. A comparison of methods for differential expression analysis of RNA-seq data. BMC Bioinformatics. 2013 Mar 9;14:91. doi: 10.1186/1471-2105-14-91. PMID 23497356
- [Background] Law CW, Chen Y, Shi W, Smyth GK. voom: Precision weights unlock linear model analysis tools for RNA-seq read counts. Genome Biol. 2014 Feb 3;15(2):R29. doi: 10.1186/gb-2014-15-2-r29. PMID 24485249
- [Background] Schmader KE, Johnson GR, Saddier P, Ciarleglio M, Wang WW, Zhang JH, Chan IS, Yeh SS, Levin MJ, Harbecke RM, Oxman MN; Shingles Prevention Study Group. Effect of a zoster vaccine on herpes zoster-related interference with functional status and health-related quality-of-life measures in older adults. J Am Geriatr Soc. 2010 Sep;58(9):1634-41. doi: 10.1111/j.1532-5415.2010.03021.x. PMID 20863322
- [Background] Drolet M, Levin MJ, Schmader KE, Johnson R, Oxman MN, Patrick D, Fournier SO, Mansi JA, Brisson M. Employment related productivity loss associated with herpes zoster and postherpetic neuralgia: a 6-month prospective study. Vaccine. 2012 Mar 9;30(12):2047-50. doi: 10.1016/j.vaccine.2012.01.045. Epub 2012 Jan 28. PMID 22285632

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hepatitis C Infected Volunteers | Healthy Volunteers
Started | 0 | 14
Completed | 0 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We plan to collect and freeze all samples and then run tests on all samples at the same time. As not all samples were collected/processed, many of the assays were not yet performed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hepatitis C Infected Volunteers | Healthy Volunteers | Total
Number analyzed (Participants) | 0 | 14 | 14
Age, Continuous [Mean (Full Range); unit: years] |  | 57 [53 to 64] | 57 [53 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 4 | 4
  Male |  | 10 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 2 | 2
  Not Hispanic or Latino |  | 11 | 11
  Unknown or Not Reported |  | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 1 | 1
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 5 | 5
  White |  | 6 | 6
  More than one race |  | 1 | 1
  Unknown or Not Reported |  | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 14 | 14

OUTCOME MEASURES:

1. Primary Outcome: Serum Zoster Antibody Level
Description: Serum zoster antibody level would be measured by gpELISA expressed in (units/mL)
Time Frame: 18 months
Population: Samples were collected but none were tested for antibody levels
Arm/Group | Hepatitis C Infected Volunteers | Healthy Volunteers
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Interferon Stimulated Gene (ISG) Expression
Description: Interferon stimulated gene (ISG) expression in PBMC will be expressed as fold-change (FCH) above baseline
Time Frame: 18 months
Population: Samples were collected and cryopreserved. RNA was collected for these samples and batched, but the RNA-Seq (for RNA expression measurements) was not run. The samples wee not analyzed and no assays were performed for this protocol.
Arm/Group | Hepatitis C Infected Volunteers | Healthy Volunteers
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Serum Biomarkers of Immune Activation(Expressed in%)
Description: Serum biomarkers of immune activation will be measured and expressed in percentage.
Time Frame: 18 months
Population: Samples were not analyzed and no assays were performed for this protocol.
Arm/Group | Hepatitis C Infected Volunteers | Healthy Volunteers
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Responder Cell Frequency
Description: Responder cell frequency: VZV specific CD4+ T cells post-vaccination (expressed in %)
Time Frame: 18 months
Population: Samples were not analyzed and no assays were performed for this protocol.
Arm/Group | Hepatitis C Infected Volunteers | Healthy Volunteers
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Interferon-gamma Response
Description: Interferon-gamma response: by ELIspot expressed as number of spot-forming cells per million PBMCs
Time Frame: 18 months
Population: Samples were not analyzed and no assays were performed for this protocol.
Arm/Group | Hepatitis C Infected Volunteers | Healthy Volunteers
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 22 months
Description: The number of participants at risk in the Hepatitis C Infected Volunteers group is zero as we didn't enroll any volunteers in that arm of the study and the study is now closed for enrollment.
Arm/Group | Hepatitis C Infected Volunteers | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/14
Other Adverse Events (participants affected / at risk) | 0/0 | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hepatitis C Infected Volunteers (N=0) | Healthy Volunteers (N=14)
Dyspnea (Cardiac disorders) | 0 (0) | 1 (1) — The incident of dyspenia occurred during the screening visits prior to receipt of the Zoster vaccine. Not related to the test article.
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) — This volunteer has a history of previously uncontrolled hypertension of several years,with a recent history of intermittent dyspnea on exertion.He had a cardiac catheterization performed prior to the administration of Zoster vaccine in this study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hepatitis C Infected Volunteers (N=0) | Healthy Volunteers (N=14)
Mild Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — The decrease in the hemoglobin level not believed to be related to the administration of the Zoster vaccine.
Mild Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — This volunteer has had intermittent chronic back pain for the past 10 years and takes Baclofen 10 mg po h.s. for pain relief. Use of Baclofen was during the screening period prior to the administration of the Zoster vaccine and therefore not related.
Dental Filling Fell Out (Gastrointestinal disorders) | 0 (0) | 1 (1) — The volunteer had a dental filling that fell out which caused a moderate amount of dental pain (one month after administration of Zoster vaccination).
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) — This episode was precipitated by psychosocial stressors at home. He has a history of bipolar disorder.
Lightheadedness (General disorders) | 0 (0) | 1 (1) — Zoster vaccination was given on 8/8/16 and lightheadedness occurred on 8/11/16.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT02590068/Prot_SAP_000.pdf